CLINICAL TRIAL: NCT07295561
Title: Salvage Surgery in Recurrent Hypopharyngeal Carcinoma: Anobservational Single-institutional Study From 1998
Brief Title: Salvage Surgery in Recurrent Hypopharyngeal Carcinoma: an Observational Single-institutional Study From 1998
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Simone Mauramati, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: Salvage_reconstruction
Record Dates: First submitted 2025-12-03; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-08

CONDITIONS: Hypopharyngeal Carcinoma
MeSH Terms: conditions — Hypopharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study will be to assess the association between the type of a surgical flap and post-operative complication in patients with hypopharyngeal cancer undergoing salvage surgery (SS) and reconstruction with free or pedicled flaps.

DETAILED DESCRIPTION:
Squamous cell carcinoma of the hypopharynx (HPSCC) is a rare but aggressive cancer, accounting for only 3-5% of all head and neck cancers. It occurs in the III-IV stage in about 60-85 % of cases, with 5-year overall survival (OS) ranging from 25 to 41%. It tends to spread in local submucosa, with an early involvement of the larynx and the locoregional tissue. Disease recurrence is around 15% to 40%, depending on the casuistry, the type of primary treatment (surgery vs. organ preservation protocols) and personal experience of each center. In recurrence setting, where indicated, salvage surgery (SS) remains the gold standard with the highest survival rates compared to conservative therapy. Generally patients are frail, with poor performance status and countless comorbidities and between 33% to 66% of cases are eligible to surgery with curative intent. In fact, in salvage setting the risk of peri-operative mortality is higher, postoperative complications are more frequent and hospital stay is longer.

Therefore, a careful selection of candidates is imperative and based on the following criteria: age and comorbidities, site of recurrence, stage, time interval since the first treatment and type of previous therapies

ELIGIBILITY:
Inclusion Criteria:

* recurrence of hypopharynx/hypopharyngolarynx cancer after the first hypopharynx/hypopharyngolarynx tumor;
* treatment with salvage surgery and reconstruction using free or pedicled flaps.

Exclusion Criteria:

* recurrence of cancer in a location other than the hypopharynx/hypopharyngolarynx or with the first tumor in a location other than the hypopharynx/hypopharyngolarynx;
* treatment with salvage surgery without flap reconstruction or with salvage treatment not involving flap reconstruction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with recurrence of hypopharynx/hypopharyngolarynx cancer after salvage surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2027-03-18 (Estimated); Study Completion 2027-03-18 (Estimated)

PRIMARY OUTCOMES:
the difference in proportions of non necrotic complications in the two groups of patients. | up to 24 months

SECONDARY OUTCOMES:
the difference in proportions of necrotic complications in the two groups of patients. | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy